CLINICAL TRIAL: NCT01704573
Title: Nicotinic Receptor Availability in Slow and Fast Nicotine Metabolizers
Brief Title: Nicotinic Receptor Levels After Stopping Smoking
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 812051; P50CA143187 (NIH)
Record Dates: First submitted 2012-10-02; First posted 2012-10-11 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Nicotine Addiction
Keywords: PET Scan
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two saliva samples will be collected at the medical screening session. A 6ml saliva sample will be used for nicotine metabolite ratio (NMR) estimation, and a 2ml saliva sample for DNA extraction (using an Oragene collection kit).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NMR by abstinence status: This study uses a mixed design with one between-subject factor (NMR: continuous variable) and one within-subject factor (session: 24 hours abstinent vs. smoking as usual) to examine NMR by abstinence status interactions on α4β2* nAChR availability using 2-[18F]-fluro-3-[2(S)-2-azethidinylmethoxy]-pyridine (2-[18F]FA) PET imaging.
  Subjects will participate in two one-hour PET sessions: a) after smoking as usual (smoking exposure standardized) and b) the other following 24 hours of smoking abstinence.
  All participants who complete both PET scans will also complete an anatomical MRI scan.
  Interventions: Drug: 2-[18F]-fluro-3-[2(S)-2-azethidinylmethoxy]-pyridine

INTERVENTIONS:
Drug: 2-[18F]-fluro-3-[2(S)-2-azethidinylmethoxy]-pyridine — The study will be performed using an Investigational New Drug (IND) Application for the 2-[18F]FA radioligand. The 2-[18F]FA radiotracer allows us to measure nicotine receptors. The PET imaging technique used at these sessions allows us to measure the amount of light that 2-[18F]FA gives off in different regions of the brain, we can estimate how many nicotine receptors are in that region.
  2-[18F]FA (radiotracer) is investigational, which means it is not approved by the United States Food and Drug Administration (FDA) for the way that it is being used in this research study. For this reason, we have received approval for all procedures in the current study including the use of 2-[18F]FA from the FDA.
  Other Names: 2-[18F]FA, 2-FA

SUMMARY:
This positron emission tomography (PET) study examines the effects of 24 hours abstinence from smoking on return to availability of neuronal nicotinic receptors in slow and fast metabolizers of nicotine.

DETAILED DESCRIPTION:
The nicotine metabolite ratio (NMR), a stable marker of nicotine clearance rate, is a robust predictor of smoking relapse. Individuals who are fast nicotine metabolizers have higher rates of relapse, compared to slow metabolizers, on nicotine replacement or placebo treatment. Nicotine exerts its reinforcing properties, in part, by binding to α4β2* nicotinic acetylcholine receptors (nAChRs) in the brain. The α4β2* nAChRs are abundant and have high affinity for nicotine relative to other nAChR subtypes. The goal of this project is to identify abstinence-induced changes in neuronal nicotinic receptor availability that may underlie risk for smoking relapse.

The investigators propose to utilize positron emission tomography (PET) imaging to examine the association of variation in nicotine metabolism with return to availability of α4β2* nAChRs during early abstinence. The investigators will measure α4β2* receptor availability using the PET radio-ligand 2-[18F]FA, administered with bolus injection, on two separate occasions: during smoking as usual and after 24 hours of abstinence. The proposed study will help us understand the neurochemical mechanisms that underlie the higher risk of relapse among faster nicotine metabolizers, thereby pointing to potential targets for tailored therapy for these smokers at increased risk.

In addition, the investigators will invite six subjects who have completed the two PET scans described above to complete a third PET scan. During this third PET scan, the investigators plan to measure α4β2* receptor availability using the PET radio-ligand 2-[18F]FA, administered as bolus plus constant infusion after 24 hours of abstinence. The purpose will be to compare α4β2* nAChR binding potential data from the bolus 2-[18F]FA infusion protocol used in the main study to the bolus plus constant infusion protocol used in this third PET scan.

The protocol of this third PET scan will help the investigators demonstrate the feasibility at the University of Pennsylvania of administering the radiotracer as a bolus plus constant infusion, and the feasibility of scanning for two hours (versus one hour in the current protocol) paradigm. This data is important pilot data for future NIH grant submissions using this radiotracer.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 65 years old.
2. Smoke 10 cigarettes per day for the previous 6 months.
3. Weigh less than 300lbs (due to limitations of the PET and MRI scanners).

Exclusion Criteria:

1. Smoking behavior:

   1. Current enrollment or plans to enroll in a smoking cessation program, or use other smoking cessation medications in the next 2 months.
   2. Provide a CO reading of less than 10 ppm at medical screening.
2. Alcohol/Drugs:

   1. History of substance abuse and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants).
   2. Positive drug screen at any of the sessions (see page 8 for list of drugs and/or contra-indicated medications).
   3. Current alcohol consumption that exceeds 25 standard drinks/week.
   4. Providing a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 at any session.
3. Medical:

   1. Women who are pregnant, planning a pregnancy, or lactating; all female subjects shall undergo a serum pregnancy test at the medical screening session and urine pregnancy tests at the two PET scans and MRI scan.
   2. Women of child-bearing age must agree in writing to use an approved method of contraception or agree to abstain from sexual intercourse
   3. History or current diagnosis of the following psychiatric diagnoses identified by the MINI (Mini International Neuropsychiatric Interview) such as psychosis, bipolar disorder, schizophrenia, major current depression, or any Axis 1 disorder
   4. Self-report of serious or unstable disease within the past 6 months (e.g., cancer [except melanoma], HIV/AIDS, stroke, angina, coronary disease, heart attack).
   5. History of epilepsy or a seizure disorder.
   6. Any medical or neurological condition that might interfere with the distribution of the radiotracer as determined by the study M.D.
4. Medication:

   a. Current use or recent discontinuation (within last 14-days) of the following medications:
   * Any form of smoking cessation medication (Zyban, Wellbutrin, Wellbutrin SR, Chantix, NRT);
   * Recent (within last 14 days) or planned use of psychotropic medications (anti-psychotics, anti-depressants, anti-anxiety, anti-panic medications, mood stabilizers, opioids, and stimulants).
   * Participants shall be instructed to refrain from using any study prohibited drugs (note - participants are allowed to take prescription medicines not in the exclusion list) throughout their participation in the study.
5. Imaging-Related Exclusion Criteria:

   1. Self-reported history of head trauma or brain (or CNS) tumor.
   2. Self-reported history of claustrophobia (contraindicated for PET and MRI).
   3. Having a cochlear implant or wearing bilateral hearing aids.
   4. Self-reported use of pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for MRI.
   5. History of gunshot wound.
   6. Circumstances or conditions that may interfere with magnetic resonance imaging (MRI)
   7. Inability to complete the baseline study procedures within four hours and/or correctly, as determined by the PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 adult, non-treatment seeking smokers, reporting consumption of greater than/equal to 10 cigarettes per day for at least 6 months will be the target population for the study. Participants will first be screened over the phone and then complete an in-person medical screen to ensure final eligibility. Enrolled participants will complete 2 PET scans and an MRI scan.
  6 smokers who have completed the study and have agreed to be re-contacted for future studies will be invited to participate in an additional procedure. Participants will be screened over the phone and complete an in-person medical screen to ensure final eligibility. Enrolled participants will complete 1 PET scan.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in α4β2* nAChR binding potential | Week 1 and up to Week 5
  This study uses a mixed design. A within-subject positron emission tomography (PET) study comparing α4β2* nAChR availability, using 2-[18F]FA PET imaging, at two timepoints (1) during smoking as usual; and (2) after 24 hours of overnight abstinence. The order of the PET scans will be counterbalanced across subjects to prevent order effects that could bias the study results. Nicotine metabolite ratio (NMR) serves as the between-subject factor.
  The minimum amount of time between scans will be separated by one week. The maximum amount of time allowable between scans will be 4 weeks.

SECONDARY OUTCOMES:
Cigarette craving | Week 0, Week 1, and up to Week 5
  The 10-item brief QSU (QSU-B) questionnaire will be used to assess smoking urges at medical screening and at each PET scanning session. The QSU contains 2 subscales (anticipation of reward, relief from negative affect).
  During each PET scanning session, the measure will be administered both before and after the PET scan.
Behavioral Performance on cognitive tasks | Week 1 and up to Week 5
  Explore potential correlations between α4β2* nAChR availability (smoking versus abstinence) with cognitive performance using 3 computer tasks: an N-back task assessing working memory, a continuous performance task assessing sustained attention, and a task assessing attentional bias to smoking cues.

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CIRNA website — http://www.med.upenn.edu/cirna/